CLINICAL TRIAL: NCT06146933
Title: Evaluierung Der Systemgenauigkeit Des Blutglucosemonitoring Systems GL22 gemäß DIN EN ISO 15197:2015.
Brief Title: System Accuracy of BGM GL22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Responsible Party: Principal Investigator, Matthes Kenning, Dr. Kerstin Rebrin, Institut fur Diabetes Karlsburg GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023_004
Record Dates: First submitted 2023-09-07; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject glucometer measurement (Experimental)
  Interventions: Diagnostic Test: Glucometer Test; Diagnostic Test: Refernce Measurement

INTERVENTIONS:
Diagnostic Test: Glucometer Test — blood glucose measurement using finger tip capillary blood using BGM
Diagnostic Test: Refernce Measurement — blood glucose measurement using finger tip capillary blood using reference method

SUMMARY:
This study assesses the system accuracy of a blood glucose monitoring system pursuant to ISO 15197

ELIGIBILITY:
Inclusion criteria:

* Male or female patients with hypo-, eu- or hyperglycaemia
* The written informed consent had to be signed
* The volunteers must be older than 18 years
* The volunteers have legal capacity and are able to understand meaning, nature and possible consequences of the procedures involved

Exclusion criteria:

* Pregnancy or lactation
* Acute or chronic diseases with the risk of aggravation by the measure
* A current constitution that does not allow participating in the study
* Participation in another study or activity with the blood glucose measuring system evaluated in the present study
* Application of substances listed in Appendix A of DIN EN ISO 15197:2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy based on DIN EN ISO 15197 | Day 1
  Assessment of the analytical measurement performance of the blood glucose monitor

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Rebrin, PhD, Study Director — Institut fur Diabetes Karlsburg GmbH
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No